CLINICAL TRIAL: NCT06065033
Title: Exercise as a Therapeutic for Those Diagnosed With Post-acute Sequelae of Covid-19
Brief Title: Exercise Interventions in Post-acute Sequelae of Covid-19
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Personnel issues.
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Siddartha Angadi, Principal Investigator, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HSR230278
Record Dates: First submitted 2023-09-29; First posted 2023-10-03 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Our approach will consist of a randomized, blinded, 2-arm, parallel-group design
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded to subject allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): Patients will perform 5 days of supervised stationary cycling exercise (with EKG telemetry) per week over a period of 4 weeks. Training heart rates will be determined based on the pre-testing VO2peak and peak heart rate (PHR).
  * Of the 5 sessions, 3 will be HIIT sessions and 2 will be MOD sessions.
  * Subjects exercising on the HIIT day will start with eight intervals of 2-min duration at 80-85% of PHR, separated by 2 min of recovery at 50% of PHR, progressing to four, 4-min intervals at 90-95% PHR, separated by 3 min at 50% PHR by the end of week 2.
  * Subjects exercising on the MOD days will perform uninterrupted for 40 minutes duration at 60-65% of PHR progressing to 40 minutes duration at 70-75% of PHR by the end of week 2.
  * Each training session will begin with a 10-min warm-up at 50% PHR and end with a 5-min cool down at 50% PHR. Exercise progression may have to be modified according to individual subject exercise tolerance.
  Interventions: Behavioral: Exercise
- Control (No Intervention): The control protocol will include a combination of light stretching and controlled breathing.

INTERVENTIONS:
Behavioral: Exercise — Patients will perform 5 days of supervised stationary cycling exercise (with EKG telemetry) per week over a period of 4 weeks. Training heart rates will be determined based on the pre-testing VO2peak and peak heart rate (PHR).
  * Of the 5 sessions, 3 will be HIIT sessions and 2 will be MOD sessions.
  * Subjects exercising on the HIIT day will start with eight intervals of 2-min duration at 80-85% of PHR, separated by 2 min of recovery at 50% of PHR, progressing to four, 4-min intervals at 90-95% PHR, separated by 3 min at 50% PHR by the end of week 2.
  * Subjects exercising on the MOD days will perform uninterrupted for 40 minutes duration at 60-65% of PHR progressing to 40 minutes duration at 70-75% of PHR by the end of week 2.
  * Each training session will begin with a 10-min warm-up at 50% PHR and end with a 5-min cool down at 50% PHR. Exercise progression may have to be modified according to individual subject exercise tolerance.
  Arms: Exercise

SUMMARY:
The COVID-19 pandemic severely impacted the medical system both directly but also through incomplete recovery from the virus in the form of post-acute sequelae of COVID-19 (PASC). PASC affects at least 9.6 million individuals as of May 2022 and continues to affect many more. PASC is a multisystem disorder often presenting with mental fog, dyspnea on exertion, and fatigue among other symptoms. The etiology of PASC is uncertain but theories include direct cytotoxicity, dysregulated immune responses, endotheliitis associated with microthrombi, eNOS uncoupling, and myocardial fibrosis with impaired ventricular compliance. To date, there are no established treatments. Exercise has the potential as a therapeutic option to improve VO2peak and improve each of the aforementioned underlying etiologies. The investigators plan to examine the effect of High-Intensity Interval Training (HIIT) and Moderate intensity exercise training (MOD) on the symptoms and exercise tolerance of patients with PASC.

The investigators approach will consist of a randomized, blinded, 2-arm, parallel-group design. Enrolled subjects will be randomly assigned to one of two groups in a 1:1 allocation ratio. All groups will undergo a 4-week intervention of 3 days of HIIT per week and 2 days of MOD per week or control of light stretching and controlled breathing. Subjects will be assessed before and after the 4-week intervention to examine the extent to which 4 weeks of the HIIT and MOD combination improves VO2peak and left ventricular diastolic function, global longitudinal strain (GLS), and global circumferential strain (GCS). Further, the investigators will explore changes in markers such as heart rate, heart rhythm, blood pressure, quality of life, exercise tolerance, and PASC symptoms as well as blood/serum markers.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years of age
* Diagnosed with Post Acute Sequelae of COVID-19
* Physician clearance to undergo exercise training (see section titled cardiorespiratory fitness testing for details; page 6)
* Complete COVID-19 vaccination status

Exclusion Criteria:

* Unstable angina or myocardial infarction in the past 4 weeks
* Uncompensated heart failure
* NYHA class IV symptoms
* Complex ventricular arrhythmias
* Musculoskeletal contraindications to stationary bicycling exercise
* Symptomatic severe aortic stenosis
* Acute pulmonary embolus
* Acute myocarditis
* Uncontrolled Hypertension as defined as systolic blood pressure > 180 mm Hg or diastolic blood pressure > 120 mm Hg
* Medication non-compliance
* Pregnant women-self reported
* COPD GOLD stage D
* Malignancy currently actively being treated
* Uncontrolled Asthma
* Uncompensated Cirrhosis of the Liver
* Chronic Kidney disease requiring dialysis therapy
* Symptomatic Anemia
* Hemoglobin <7g/dL
* Poorly controlled diabetes or A1c>9%
* BMI >35kg/m2
* Pulmonary Hypertension stage IV
* Any condition requiring supplemental oxygen
* Multiple Sclerosis

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09-09 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-03-29 (Actual)

PRIMARY OUTCOMES:
VO2peak | 4 weeks
  Change in VO2peak (L/min) measured pre- and post-intervention
Left ventricular strain | 4 weeks
  Global longitudinal strain and global circumferential strain measured pre- and post-intervention
Left ventricular diastolic function | 4 weeks
  Diastolic dysfunction grade measured pre- and post-intervention

SECONDARY OUTCOMES:
Forced expiratory volume in one second (FEV1) | 4 weeks
  FEV1 measured via spirometry pre- and post-intervention
Forced vital capacity (FVC) | 4 weeks
  FVC measured via spirometry pre- and post-intervention
Post COVID-19 Functional Status scale | 4 weeks
  Measures subjects functional limitations due to COVID-19 and will be measured via pre- and post-intervention
Symptom Burden Questionnaire for Long Covid (SBQ-LC) | 4 weeks
  Burden of symptoms will be via the SBQ-LC measured pre- and post-intervention
International Physical Activity Questionnaire (IPAQ) | 4 weeks
  Physical activity levels will be assessed via IPAQ measured pre- and post-intervention
NTproBNP | 4 weeks
  Assess changes in NTproBNP (pg/ml) as a biomarker of myocardial strain at pre- and post-intervention
C-reactive protein (CRP) | 4 weeks
  C-reactive protein (mg/dl) will be used as a biomarker for inflammation to be measured pre- and post-intervention
Lipids | 4 weeks
  A lipid panel will be performed to measure total cholesterol, triglycerides, high-density lipoproteins, and low-density lipoprotein (mg/dl) to assess changes in cardiometabolic health pre- and post-intervention
Fasting glucose | 4 weeks
  Fasting blood glucose levels (mg/dl) will be tested to assess changes in cardiometabolic health pre- and post-intervention
Insulin | 4 weeks
  Fasting insulin levels (U/ml) will be tested to assess changes in cardiometabolic health pre- and post-intervention
Erythrocyte sedimentation rate (ESR) | 4 weeks
  ESR will be measured to assess inflammation pre- and post-intervention
IL-1 | 4 weeks
  Inflammation will be measured via IL-1 pre- and post-intervention
IL-6 | 4 weeks
  Inflammation will be measured via IL-6 pre- and post-intervention
TNF-a | 4 weeks
  Inflammation will be measured via TNF-a pre- and post-intervention
Fibrinogen | 4 weeks
  Fibrinogen will be measured pre- and post-intervention to measure clotting
D-dimer | 4 weeks
  D-dimer will be measured pre- and post-intervention to measure clotting

CONTACTS AND LOCATIONS:
Overall Officials: Siddhartha S Angadi, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia University Hospital, Charlottesville, Virginia, United States